CLINICAL TRIAL: NCT04539158
Title: Efficacy and Safety of Dual Direct Current Cardioversion Versus Single Direct Current Cardioversion as an Initial Treatment Strategy in Obese Patients
Brief Title: Single vs. Dual-DCCV in Obese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Daniel P Morin, MD MPH FHRS (Other)
Responsible Party: Sponsor-Investigator, Dr. Daniel P Morin, MD MPH FHRS, Medical Director of Cardiovascular Research, Ochsner Health System
Organization: Ochsner Health System (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2020.048
Record Dates: First submitted 2020-08-30; First posted 2020-09-04 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electric Countershock

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned in a 1:1 fashion to either single-DCCV or dual-DCCV treatment.
  All patients will have 4 defibrillation pads placed: two pads placed in the right infraclavicular and left flank regions, plus two pads placed in the left infraclavicular and right flank regions.
  Patients randomized to single-DCCV will receive a single 200J shock using the "primary" (or right anterior-left posterior) pair of pads. Patients assigned to dual-DCCV will receive two simultaneous 200J shocks (from both the "primary" and "secondary" set of defibrillator pads), totaling 400J delivered.
  Patients in the single-DCCV group whose initial shock fails to restore normal sinus rhythm will be crossed over to the dual-DCCV group. Patients in the dual-DCCV group will receive up to three attempts at DCCV, as needed, at the discretion of the attending electrophysiologist.
Who Masked: Participant
Masking Description: All patients will have 4 defibrillation pads placed: two pads placed in the right infraclavicular and left flank regions, plus two pads placed in the left infraclavicular and right flank regions. Patients will not be told which arm they are randomized to during the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- single-DCCV group (Active Comparator): Patients randomized to single-DCCV will be given a single 200J shock using the "primary" (or right anterior-left posterior) pair of pads.
  Interventions: Device: Direct Current Cardioversion
- dual-DCCV group (Experimental): Patients assigned to dual-DCCV will receive two simultaneous 200J shocks (from both the "primary" and "secondary" set of defibrillator pads), totaling 400J delivered.
  Interventions: Device: Direct Current Cardioversion

INTERVENTIONS:
Device: Direct Current Cardioversion — The patient is sedated and shocked using an external defibrillator to terminate the arrhythmia and restore a normal intrinsic rhythm (i.e., normal sinus rhythm).

SUMMARY:
Currently, the usual initial strategy for direct current cardioversion (DCCV) typically involves delivering 200J of electricity between two pads placed in the anterior and posterior positions (i.e., one on the chest and one on the back). However, this technique may be less likely to result in successful cardioversion in obese patients (BMI ≥30 kg/m2). Failure to achieve sinus rhythm then necessitates additional shocks, which still may ultimately fail to terminate the patient's atrial fibrillation, thereby increasing the likelihood of adverse events from multiple cardioversion attempts

"Dual-DCCV" is a technique in which four pads are used to deliver two simultaneous shocks of 200J, totaling 400J. Guidelines published by the American Heart Association/American College of Cardiology/Heart Rhythm Society and the European Society of Cardiology provide only general guidance regarding the appropriate technique and energy selection in patients undergoing cardioversion, with no specific recommendations pertaining to dual-DCCV or obese patients.

This study aims to assess the safety and efficacy of dual-DCCV as an initial treatment strategy, compared to standard single-DCCV, in the obese population.

DETAILED DESCRIPTION:
Patients with sustained atrial fibrillation and obesity who are scheduled for a cardioversion for atrial fibrillation will provide written informed consent prior to starting the procedure. Patients will be randomly assigned in a 1:1 fashion to either single-DCCV or dual-DCCV treatment.

All patients will have 4 defibrillation pads placed: two pads placed in the right infraclavicular region and left flank region, plus two pads placed in the left infraclavicular and right flank region.

All patients will receive moderate sedation immediately prior to and during cardioversion.

Patients randomized to single-DCCV will be given a single 200J shock using the "primary" (or right anterior-left posterior) pair of pads. Patients assigned to dual-DCCV will receive two simultaneous 200J shocks (from both the "primary" and "secondary" set of defibrillator pads), totaling 400J delivered.

Patients in the single-DCCV group whose initial shock fails to restore normal sinus rhythm will be crossed over to the dual-DCCV group. Patients in the dual-DCCV group will receive up to three attempts at DCCV, as needed, at the discretion of the attending electrophysiologist.

One hour after cardioversion is completed, patients will be asked if they experienced any chest discomfort related to cardioversion and, if applicable, will rate their chest discomfort using a pain scale from 0-10.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Atrial fibrillation (paroxysmal, persistent, and long-standing persistent)
* Obesity (defined as body mass index [BMI] ≥35 kg/m2). Of note, our current institutional protocol uses weight >250 lbs as an indication for dual-DCCV. An average height of 70 inches equates to BMI ~35 kg/m2
* Adequate anticoagulation at the time of the cardioversion (one of the following):

  * Coumadin with an INR >2
  * Direct oral anticoagulants (apixaban, dabigatran, rivaroxaban, or edoxaban)
  * Subcutaneous low molecular-weight heparin or IV unfractionated heparin
* If the duration of atrial fibrillation is >48 hours (or unknown): trans-esophageal echocardiography (TEE) performed prior to cardioversion to document the absence of a left atrial thrombus, or continuous therapeutic anticoagulation for a minimum of 3 weeks prior to cardioversion
* Able to maintain uninterrupted therapeutic anticoagulation after cardioversion, for at least one month

Exclusion Criteria:

* Contraindication to cardioversion
* Not on adequate anticoagulation
* Emergent cardioversion
* Incarceration
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Successful return to sinus rhythm confirmed via rhythm strip ECG (regardless of duration) immediately following DCCV | 0-1 hours
  Participant cardiac rhythm verified to have returned to sinus rhythm by single-lead rhythm strip ECG obtained via the defibrillator device.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel P Morin, MD, Principal Investigator — Ochsner Health System
Locations (3):
- United States (3):
  - Ochsner Medical Center - West Bank, Gretna, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - LSU Health Sciences Center - Shreveport, Shreveport, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gallagher MM, Guo XH, Poloniecki JD, Guan Yap Y, Ward D, Camm AJ. Initial energy setting, outcome and efficiency in direct current cardioversion of atrial fibrillation and flutter. J Am Coll Cardiol. 2001 Nov 1;38(5):1498-504. doi: 10.1016/s0735-1097(01)01540-6. PMID 11691530
- [Background] Gardner MW, Yadava M, Raitt MH, Elman MR, Zarraga IG, MacMurdy KS, Dalouk KA, Jessel PM. Effectiveness of dual external direct current cardioversion for initial cardioversion in atrial fibrillation. J Cardiovasc Electrophysiol. 2019 Sep;30(9):1636-1643. doi: 10.1111/jce.13994. Epub 2019 Jun 11. PMID 31111594
- [Background] Glover BM, Walsh SJ, McCann CJ, Moore MJ, Manoharan G, Dalzell GW, McAllister A, McClements B, McEneaney DJ, Trouton TG, Mathew TP, Adgey AA. Biphasic energy selection for transthoracic cardioversion of atrial fibrillation. The BEST AF Trial. Heart. 2008 Jul;94(7):884-7. doi: 10.1136/hrt.2007.120782. Epub 2007 Jun 25. PMID 17591649
- [Background] Gurevitz OT, Ammash NM, Malouf JF, Chandrasekaran K, Rosales AG, Ballman KV, Hammill SC, White RD, Gersh BJ, Friedman PA. Comparative efficacy of monophasic and biphasic waveforms for transthoracic cardioversion of atrial fibrillation and atrial flutter. Am Heart J. 2005 Feb;149(2):316-21. doi: 10.1016/j.ahj.2004.07.007. PMID 15846271
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- [Background] Kirchhof P, Andresen D, Bosch R, Borggrefe M, Meinertz T, Parade U, Ravens U, Samol A, Steinbeck G, Treszl A, Wegscheider K, Breithardt G. Short-term versus long-term antiarrhythmic drug treatment after cardioversion of atrial fibrillation (Flec-SL): a prospective, randomised, open-label, blinded endpoint assessment trial. Lancet. 2012 Jul 21;380(9838):238-46. doi: 10.1016/S0140-6736(12)60570-4. Epub 2012 Jun 18. PMID 22713626
- [Background] Levy S, Lauribe P, Dolla E, Kou W, Kadish A, Calkins H, Pagannelli F, Moyal C, Bremondy M, Schork A, et al. A randomized comparison of external and internal cardioversion of chronic atrial fibrillation. Circulation. 1992 Nov;86(5):1415-20. doi: 10.1161/01.cir.86.5.1415. PMID 1423954
- [Background] Mittal S, Ayati S, Stein KM, Schwartzman D, Cavlovich D, Tchou PJ, Markowitz SM, Slotwiner DJ, Scheiner MA, Lerman BB. Transthoracic cardioversion of atrial fibrillation: comparison of rectilinear biphasic versus damped sine wave monophasic shocks. Circulation. 2000 Mar 21;101(11):1282-7. doi: 10.1161/01.cir.101.11.1282. PMID 10725288
- [Background] Oral H, Souza JJ, Michaud GF, Knight BP, Goyal R, Strickberger SA, Morady F. Facilitating transthoracic cardioversion of atrial fibrillation with ibutilide pretreatment. N Engl J Med. 1999 Jun 17;340(24):1849-54. doi: 10.1056/NEJM199906173402401. PMID 10369847
- [Background] Schmidt AS, Lauridsen KG, Torp P, Bach LF, Rickers H, Lofgren B. Maximum-fixed energy shocks for cardioverting atrial fibrillation. Eur Heart J. 2020 Feb 1;41(5):626-631. doi: 10.1093/eurheartj/ehz585. PMID 31504412
- [Background] Shelton RJ, Brown BD, Allinson A, Johnson T, Smales C, Jolly S, Cleland JG. A comparison between monophasic and biphasic defibrillation for the cardioversion of persistent atrial fibrillation in patients with and without heart failure. Int J Cardiol. 2011 Mar 17;147(3):405-8. doi: 10.1016/j.ijcard.2009.09.545. Epub 2009 Oct 25. PMID 19861229
- [Background] Voskoboinik A, Moskovitch J, Plunkett G, Bloom J, Wong G, Nalliah C, Prabhu S, Sugumar H, Paramasweran R, McLellan A, Ling LH, Goh CY, Noaman S, Fernando H, Wong M, Taylor AJ, Kalman JM, Kistler PM. Cardioversion of atrial fibrillation in obese patients: Results from the Cardioversion-BMI randomized controlled trial. J Cardiovasc Electrophysiol. 2019 Feb;30(2):155-161. doi: 10.1111/jce.13786. Epub 2018 Nov 14. PMID 30375104
- [Derived] Aymond JD, Sanchez AM, Castine MR, Bernard ML, Khatib S, Hiltbold AE, Polin GM, Rogers PA, Dominic PS, Velasco-Gonzalez C, Morin DP. Dual vs Single Cardioversion of Atrial Fibrillation in Patients With Obesity: A Randomized Clinical Trial. JAMA Cardiol. 2024 Jul 1;9(7):641-648. doi: 10.1001/jamacardio.2024.1091. PMID 38776097